CLINICAL TRIAL: NCT02614638
Title: Evaluation of the Impact of the Presence of a Pharmacy Technician on the Quality and Cost of Drug Therapy in the Hepato-Gastroenterology Department of the Nîmes University Hospital
Brief Title: Evaluation of the Impact of the Presence of a Pharmacy Technician on the Quality and Cost of Drug Therapy
Acronym: OPTI-PP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: LOCAL/2015/GL-01; 2015-A01309-40 (Other: RCB number)
Record Dates: First submitted 2015-11-19; First posted 2015-11-25 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2017-01

CONDITIONS: Hospitalization

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1st observational period (before experimental intervention) (Active Comparator): Patients in this arm are included during a first month of observation before the intervention is implemented.
  Intervention: One month of department-wide observation
  Interventions: Other: One month of department-wide observation
- 2nd obs. period (during experimental intervention) (Experimental): Following a one-month wash-out period, patients in this arm are included during a second month of observation during which the intervention is implemented.
  Intervention: Pharm Tech participates in department
  Interventions: Other: Pharm Tech participates in department

INTERVENTIONS:
Other: One month of department-wide observation — A pharmacy technician will be present full time in the care unit from Monday to Friday between 8:30 and 17h for 1 month for observational purposes only. During this phase, the pharmacy technician observes the current practices of preparation and administration of medication by nurses. He / she will collect medication errors and other observational data.
  Arms: 1st observational period (before experimental intervention)
Other: Pharm Tech participates in department — Following a 1 month wash-out period, a pharmacy technician will again be present full time (in practice, two technicians will relay each other) in the care unit from Monday to Friday between 8:30 and 17h for 1 month. He/she will actively take part in drug care activities in the department: management of product pathways, verification of injectable preparation, advice, etc. Medication errors and other observational data will be collected.
  Arms: 2nd obs. period (during experimental intervention)

SUMMARY:
The main objective of this study is to evaluate the impact of the presence of a pharmacy technician in a care unit (Hepato-Gastroenterology Department) on detected medication errors.

This is a before-after study consisting of three sequential phases:

Month 1: one month of observation of what is happening in the department Month 2: one month wash out period Month 3: active participation of a pharmacy technician in the department

DETAILED DESCRIPTION:
The secondary objectives of this study are:

A- To assess the impact of the presence of a pharmacy technician on the ratio of the number of patients with at least one medication error / number of included patients hospitalized in the service.

B- To characterize detected medication errors.

C- To identify and evaluate the potential causes of medication errors.

D- To evaluate whether the presence of a pharmacy technician reduces nursing time spent on medication management.

E- To evaluate the economic impact of the presence of a pharmacy technician.

F- To evaluate the acceptability of the intervention by the nursing staff and pharmacy technicians using questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* The patient must be insured or beneficiary of a health insurance plan
* The patient is hospitalized in the Hepato-Gastroenterology Department of the Nîmes University Hospital

Exclusion Criteria:

* The patient is under judicial protection
* The patient, or his/her legal guardian, expresses opposition to participation in the study
* It is impossible to correctly inform the patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2016-09; Primary Completion 2016-12-16 (Actual); Study Completion 2016-12-16 (Actual)

PRIMARY OUTCOMES:
The following ratio (relative units): Number of medication errors / number of medications administered and omitted from among all those listed on the prescription for admission | 5 days
  Primary Outcome Measure as given in protocol: Number of medication errors / number of medications administered and omitted from among all those listed on the prescription for admission (during month 1 versus during month 3).

SECONDARY OUTCOMES:
Number of patients with at least one medication error / total number of hospitalized patients included in the service | 5 days
For each medication error: the name of the drug | 5 days
For each medication error: the type of error | 5 days
  Errors are classifies as one of the following types:
  Omission; Drug; Dosage form; Expired or damaged drug; Dose; Concentration; Frequency of administration; Administration technique; Route of Administration; Rate of administration; Duration of administration; Administration Time; Patient; Drug interaction.
For each medication error: the severity index | 5 days
For each medication error: when (which step) the error occurred during the drug pathway | 5 days
  The considered steps are:
  Writing the prescription Medical decision for the prescription Transcription Pharmaceutical analysis Deliverance Preparation / reconstitution Pillbox Administration Procurement Storage Compliance Therapeutic and clinical follow-up
For each medication error: the evolution of the adverse drug event, if occurred | 5 days
For each medication error: the criticality of the error | 5 days
  Criticality is graded according to the following classes:
  1. C: no potential harm to the patient;
  2. D: treatment or increased monitoring without harm to the patient
  3. (E to I): potential harm to the patient
  3E: treatment or surgery with temporary harm 3F: longer duration of hospitalization with temporary harm 3G: permanent harm 3H: involving a life-threatening harm 3I: death
  Criticality is determined by the concordance of two, independent expert opinions; or, in case of discordance, the concordance of 2 out 3 expert opinions.
The potential causes of medication errors | 5 days
The average number of interruptions per hour during preparation or administration of drug doses by nurses | 5 days
The number of patients for whom personal treatments were managed by the nursing staff on admission / number of patients who brought their personal treatments to the care unit | 5 days
The number of patients for whom personal treatments were returned by the nursing staff at hospital discharge / number of patients who brought their personal treatments to the care unit | 5 days
Nursing staff time dedicated to: the preparation of individual doses | 5 days
Nursing staff time dedicated to: ordering health products | 5 days
Nursing staff time dedicated to: stock management and exceptional orders | 5 days
Nursing staff time dedicated to: the delivery, receipt and storage of health products | 5 days
Nursing staff time dedicated to: cabinet inventories | 5 days
Nursing staff time dedicated to: the management of expired drugs | 5 days
The number of calls made to the central pharmacy | 5 days
Staff time dedicated to managing exceptional requests | 5 days
The number of drugs consumed | 5 days
The number of medical devices consumed | 5 days
The number of immobilized drugs | 5 days
The number of immobilized medical devices | 5 days
The cost of adverse drug events care | 5 days
Care staff satisfaction questionnaire | 5 days
Pharmacy technician satisfaction questionnaire | 5 days

CONTACTS AND LOCATIONS:
Overall Officials: Géraldine Leguelinel-Blache, PharmD, PhD, Study Director — Centre Hospitalier Universitaire de Nîmes
Locations (1):
- CHRU de Nîmes - Hôpital Universitaire Carémeau, Nîmes, France